CLINICAL TRIAL: NCT05226806
Title: Connect2Move: Valorization of Natural Cardio Trekking Hiking Trails Through Open Innovation for the Sustainable Promotion of Health-oriented Tourism Across Generations
Brief Title: Connect2Move: Valorization of Natural Cardio Trekking Hiking Trails
Acronym: Connect2Move
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Ludwig Boltzmann Institute for Digital Health and Prevention (Other); Paracelsus Medical University (Other); Salzburg Research Forschungsgesellschaft mbH (Unknown); Klinik St. Irmingard - Fachklinik für Onkologie, Kardiologie, Psychosomatik und Psychotraumatologie (Unknown)
Responsible Party: Sponsor
Other Study IDs: 527/20 S; AB296 (Other Grant/Funding Number: INTERREG Bavaria-Austria 2014-2020, EU Regional Development)
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2022-01

CONDITIONS: Cardiovascular Prevention; Healthy; Healthy Lifestyle
Keywords: Cardioresipratory fitness; Hiking; Cardiovascular prevention; Exercise; Outdoor sports
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Inclusion criteria: both, mals and female, age 45 years and older. Exclusion criteria: Medical contraindications for a maximum stress test and endurance test by the attending physician
  Pathologies in the context of the preliminary examinations:
  * Acute and chronic cardiovascular diseases except arterial hypertension (systolic blood pressure ≥140 mmHg and diastolic blood pressure ≥90 mmHg in untreated and drug-treated participants) and minor valve insufficiency
  * Acute and chronic lung diseases
  * Liver and kidney diseases
  * diabetes mellitus
  * Alcohol (> 30g / day) or drug abuse
  * Obesity from grade 2 (body mass index> 35 kg / m²)
  * Orthopedic diseases with reduced physical performance
  * Existing pregnancy
  Interventions: Other: Measurement of cardiorespiratory performance in 3 different settings; Other: GENERAL CARDIO HIKES AS PART OF GENERAL TOURIST OFFER OF MUNICIPALITIES

INTERVENTIONS:
Other: Measurement of cardiorespiratory performance in 3 different settings — The study is divided into three examinations days, which extend over a maximum of 2 weeks:
  * Day 1: Inclusion examination, time required: 1.5 hours Taking anamnesis, medical examination and blood drawing, determination of PROCAM score, Framingham score, ESC score, anthropometric measurements, questionnaires (IPAQ-physical activity, health status / quality of life (SF 36)), pulmonary function test, resting ECG, echocardiography, heart rate variability measurement (VO2max determination), spiroergometry (modified Bruce protocol) on the treadmill incl. inquiries about the BORG scale
  * Day 2: 1 km test trail, Time required: 1 hour: Completion of a 1 km cardio test path including mobile spiroergometry
  * Day 3: 8 km hike, time required approx. 3.5 hours: Participation in a guided cardio hike over 8 km, if applicable, including spiroergometry Afterwards (In Austria only): Logging of physical activity, physical motivation and accompanying circumstances over a period of 3 weeks
Other: GENERAL CARDIO HIKES AS PART OF GENERAL TOURIST OFFER OF MUNICIPALITIES — General cardio hikes (WITHOUT spirometric breathing gas analysis) on the selected hiking trails. Measurement of the heart rate as well as the route, time and walking speed using GPS geotracking using an anonymized user profile. User survey regarding the user-friendliness of the application.

SUMMARY:
Regular exercise improves performance and reduces the risk of cardiovascular disease. Endurance and strength training are therefore forms of therapy with a high level of evidence in the prevention and rehabilitation of cardiovascular diseases. In this context, Hiking has a special role, as endurance exercise not only has a cardio-preventive effect, but also other health-promoting effects can be achieved through exercise in nature. However, intense physical activity can also trigger cardiovascular events, especially in poorly trained people. Hiking shows a particularly high rate of cardiovascular events including death. In addition to the incorrect assessment of the cardiovascular risk profile and physical performance, weather conditions (temperature, wind, precipitation) are often not included in the planning, which in combination further increases the risk of accidents. Hikers are rarely aware of the increased risk and prevent it through preventive medical examinations. Heart health can be assessed through a stress test or ergometry and at the same time endurance performance can be determined in the laboratory and training recommendations can be given based on the results. In order to use hiking specifically to prevent cardiovascular diseases and to reduce the risk of hiking accidents, this study sets the following goals:

1. Development, validation and dissemination of a standardized 1km cardio trekking test trail to record the individual physical endurance performance (= cardio profile), with the aim of personal categorization / determination of the stress intensities when walking and hiking on medium-sized hiking trails and alpine pastures .
2. Scientific conception and mapping of individual cardio profile standard routes through application-based data evaluation (digital cardio profile app) of the cardio trekking test trail for hiking tours in the partner regions Werfenweng and Aschau im Chiemgau.

The implementation of these goals should not replace the medical preventive examination, but serve as an additional prevention method.

DETAILED DESCRIPTION:
This present study is part of the German Austrian Connect2Move project. The aim will be the appreciation of natural and evidence-based cardio trekking trails through open innovation methods for the sustainable promotion of cross-generational, health-oriented tourism,The project has been funded via the European Regional Development Fund "INTERREG V-A Programme Austria-Bavaria - 2014-2020" . This project aims to redesign existing hiking routes into themed trails and digitally redesign by integrating cardiovascular load (e.g. HF heart rate) next to the general description of the length, altitude, nature of the path, and duration. For valorization and implementation in the participating communities, an open innovation approach is chosen, which is supported scientifically and medically and involves regional stakeholders and the population.

Within the multicenter-exporatory study the following research aims will be adressed:

1. Development, validation and dissemination of a standardized 1km cardio trekking test trail to record the individual physical endurance performance (= cardio profile), with the aim of personal categorization / determination of the stress intensities when walking and hiking on medium-sized hiking trails and alpine pastures .
2. Scientific conception and mapping of individual cardio profile standard routes through application-based data evaluation (digital cardio profile app) of the cardio trekking test trail for hiking tours in the partner regions Werfenweng and Aschau im Chiemgau.

The implementation of these goals should not replace the medical preventive examination, but serve as an additional prevention method.

The study is divided into three examinations, which extend over a maximum of 2 weeks:

Day 1: Inclusion examination at the St. Irmingard Clinic in Prien a. Chiemsee Time required: approx. 1.5 hours

* Medical anamnesis interview
* Anthropometric studies
* Blood draw
* Resting ECG
* Cardiac ultrasound / echocardiography
* Spiroergometry on the treadmill

Day 2: 1 km test trail in Aschau i. Chiemgau Time required: approx. 1 hour

• Completion of a 1 km cardio test path including mobile spiroergometry

Day 3: 8 km hike in Aschau i. Chiemgau Time required approx. 3 hours

* Participation in a guided cardio hike over 8 km
* If applicable, including spiroergometry (according to the arrangement)

Afterwards (in Austria only) : Logging of physical activity, physical motivation and accompanying circumstances over a period of 3 weeks

The initial examinations and standardized laboratory tests are carried out for the Austrian participants at the University Institute for Sports Medicine Salzburg in cooperation with the Ludwig Boltzmann Institute for Digital Health and Prevention. The German participants will be examined in the Klinik, St. Irmingard in Prien am Chiemsee, Germany in cooperation with the Chair for Preventive Pediatrics at the Technical University of Munich.

Investigations include:

* Taking anamnesis
* medical examination
* Determination of PROCAM score, Framingham score, ESC score
* Anthropometric measurements (height, weight)
* Questionnaires (physical activity (IPAQ), health status / quality of life (SF 36))
* Pulmonary function test
* Resting ECG
* Echocardiography
* Heart rate variability measurement using Polar (VO2max determination)
* Ergospirometry (modified Bruce protocol) on the treadmill with additional inquiries about the BORG scale
* Blood drawing:

  ○ Routine parameters:
  * Small blood count
  * Blood sedimentation
  * sodium
  * potassium
  * calcium
  * Glutamate pyruvate transaminase (GPT)
  * Gamma-glutamyltransferase (ℽ-GT)
  * lactate dehydrogenase (LDH)
  * creatinine
  * uric acid
  * Creatine kinase (CK)
  * cholesterol
  * triglycerides
  * high-density lipoprotein (HDL)
  * Low-density lipoprotein (LDL)
  * Thyroid stimulating hormone (TSH)
  * glucose (sober) Explanation / issue of fitness bracelets and smartphone app for logging movement, movement motivation and accompanying circumstances over a period of 3 weeks
* Pregnancy test to rule out an existing pregnancy in women

FIELD TEST:

The field test measurements are carried out in the respective partner regions of the Interreg project. This includes a Cardio-Trekking-Test Trail (CTTT), a cardio hike. The Austrian participants will be tested in the municipality of Werfenweng, the German participants in the municipality of Aschau im Chiemgau.

CARDIO TREKKING TEST TRAIL (CTTT) Immediately after the laboratory test, the performance should be determined on a standardized 1km test route (defined route profile 1000 - max. 1500m, 0-200 meters in altitude). The subjects should cover this CTTT at a submaximal speed according to the BORG scale of 15 (strenuous).

The test subjects are equipped with a mobile spirometry (K5, Cosmed, mixed chamber) unit that measures and records respiratory volumes and gases throughout the test route. At the same time, the heart rate is recorded using a chest strap. The distance covered and the time required for this are recorded using a validated app. At the end of the examination, the participant himself exports the data from the app and sends it to the study center.

A mathematical model is created from the recorded data of the spirometry and the app, which, based on the data collected by the app, enables the study participant to derive the maximum oxygen uptake as a surrogate of the individual cardiovascular performance without the technically complex spirometry. This should enable a validated, automated and technically simple recommendation of stress intensities.

CARDIO HIKE AS PART OF CLINICAL STUDY The 72 test subjects in Austria who took part in the clinical study, as well as the 72 test subjects in Germany, hike, accompanied by the sports scientists involved, on previously selected cardio hiking trails. The selection criteria for the paths are defined in the study consortium according to tourism, sports science and medical aspects (LBI Salzburg, Salzburg Research, TUM; St. Irimingard Klinik Prien and all partners and regions) - visitor frequency, degrees of difficulty, sights, cultural heritage are taken into account.

Based on the results of the 1km test path, the participants receive recommendations as to the individual pulse ranges in which they should complete the hike in order to stay in a moderate intensity range. During the cardio hike, the heart rate, the breathing gas exchange, the length of the path, as well as the incline and the walking speed are measured using GPS tracking. The aim of this study is to collect heart rate data in relation to the distance traveled during the hike. Using the digitally supported application, the load, the walking speed and the path (including the height profiles) can be recorded. The data is recorded anonymously and is used to map the route according to the intensity of the load. At the end of the examination, the participant himself exports the data from the app and sends it to the study center.

GENERAL CARDIO HIKES AS PART OF GENERAL TOURIST OFFER OF MUNICIPALITIES In addition, general cardio hikes (WITHOUT spirometric breathing gas analysis) should take place on the selected hiking trails. There is no age limit for general cardio hikes. Only the heart rate is determined as well as the route, time and walking speed using GPS geotracking using an anonymized user profile. For the implementation of the general cardio hikes in the participating communities, training of hiking guides / sports scientists takes place in the two pilot regions on the German and Austrian side. 25 hikes with a maximum of 10 people from the general population are planned. A user survey regarding the user-friendliness of the application is planned.

ENVIRONMENTAL CONDITIONS DURING FIELD TEST In order to keep the temperature difference between the 1km field test and the spiroergometry in the laboratory as low as possible, the laboratory test is carried out at a standardized temperature of 20 ° C and thus the expected average daily temperature of the study months in the test regions. A performance-physiologically relevant influence on the heart rate response is to be expected from a temperature of 26 ° C. If this temperature is exceeded on a field test day, the 1km field test will be postponed to another day. The humidity is recorded in the field as well as in the laboratory test, and attention is paid to ensuring that the study participants are adequately hydrated.

Appropriate hiking equipment and adequate hydration are ensured on all field hikes. The field investigations are not carried out in the event of objective environmental hazards for the participants (thunderstorms, lightning strikes, mudslides, etc.).

In Austria only, a survey of physical activity, motivation to move and eating behavior in everyday life will be carried out. Within this survey the following data types are collected over a period of 3 weeks using a specially developed smartphone app :

* Survey on stress, emotions, motivation to exercise and eating in everyday life via smartphone: When participating in the study, the test subjects are asked several times a day using a specially developed smartphone application to answer various questions about their mental health and eating behavior (e.g. "How nervous and stressed are you at the moment? "," How strongly are you currently motivated for exercise and sport? "). The request for input is given by an acoustic signal.
* Smartphone data. Data on usage patterns and sensor data are stored in the background. The data processing is limited to the research questions and takes place without inexpedient techniques and data comparisons.

The following data is stored and processed: background volume; relative movement of the mobile phone (with the accelerometer and accelerometers of the smartphone); Time and duration of phone calls without storing the numbers, time of messages (e.g. SMS, WhatsApp) without collecting identifying information such as content, addresses, numbers); Screen activity (so-called touch events); Screen-On-Time (illuminated display); Ambient brightness; Data volume per unit of time (total value of all smartphone activities on the Internet); On and off times of the mobile phone.

GPS data is only used to decrypt user-defined 'zones', which you enter yourself. A maximum of three "zones" are recorded: "At home", "work / school", "hobby". The application and the server only have these three rooms available, but not the absolute GPS coordinates. Furthermore, the current weather and traffic density can be deduced from GPS coordinates, which in turn do not allow any conclusions to be drawn about absolute GPS coordinates. The translation of the GPS data into zones or weather / traffic data takes place directly on the smartphone, so GPS data is never transferred to the server.

• Data on physical activity: A commercially available portable measuring device that is made available to the test subjects at the initial examination for the duration of the study ("wearable", e.g. armband, chest strap) is used to record data on their exercise intensity and heart rate to determine the extent capture actual activity.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* Medical contraindications for a maximum stress test and endurance test by the attending physician

Pathologies in the context of the preliminary examinations:

* Acute and chronic cardiovascular diseases except arterial hypertension (systolic blood pressure ≥140 mmHg and diastolic blood pressure ≥90 mmHg in untreated and drug-treated participants) and minor valve insufficiency
* Acute and chronic lung diseases
* Liver and kidney diseases
* diabetes mellitus
* Alcohol (> 30g / day) or drug abuse
* Obesity from grade 2 (body mass index> 35 kg / m²)
* Orthopedic diseases with reduced physical performance
* Existing pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Development, validation and dissemination of a standardized 1 km Cardio-Trekking-Test Trail to record the individual physical endurance capacity | 2 days
  The primary research aim is to answer the following research question:
  Development, validation and dissemination of a standardized 1 km Cardio-Trekking-Test Trail to record the individual physical endurance capacity (= CardioProfil), with the aim of personal categorization / determination of the stress intensities when walking and hiking on medium-sized hiking trails and alpine pastures

SECONDARY OUTCOMES:
Scientific conception and mapping of cardio profile standard routes through application-based data evaluation (digital cardio profile application) of the cardio trekking test trails | 1 day
  Scientific conception and mapping of cardio profile standard routes through application-based data evaluation (digital cardio profile application) of the cardio trekking test trails for hiking routes in the partner regions Werfenweng and Aschau im Chiemgau. Tourist, sports science and medical aspects (TUM, St. Irmingard Klinik Prien, LBI and all partners and regions) such as visitor frequency, degree of difficulty, sights and cultural heritage are also included as selection criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Technical University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eisenberger L, Mayr B, Beck M, Venek V, Kranzinger C, Menzl A, Jahn I, Sareban M, Oberhoffer-Fritz R, Niebauer J, Bohm B. Assessment of Exercise Intensity for Uphill Walking in Healthy Adults Performed Indoors and Outdoors. Int J Environ Res Public Health. 2022 Dec 12;19(24):16662. doi: 10.3390/ijerph192416662. PMID 36554543
- [Derived] Mayr B, Beck M, Eisenberger L, Venek V, Kranzinger C, Menzl A, Reich B, Hornung-Prahauser V, Oberhoffer-Fritz R, Bohm B, Niebauer J. Valorization of Natural Cardio Trekking Trails Through Open Innovation for the Promotion of Sustainable Cross-generational Health-Oriented Tourism in the Connect2Move Project: Protocol for a Cross-sectional Study. JMIR Res Protoc. 2022 Jul 13;11(7):e39038. doi: 10.2196/39038. PMID 35830223
- See also: Study and project website (in German only) — https://connect2move-wandern.eu/